CLINICAL TRIAL: NCT01639729
Title: Effect of Delivery Route on the Pharmacokinetics of Sufentanil NanoTab® in Healthy Subjects
Brief Title: Effect of Delivery Route on PK of Sufentanil NanoTab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IAP102
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Results first posted 2014-05-21 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Pharmacokinetics
Keywords: pharmacokinetics; area under curve; time to maximum concentration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 - Treatment A, B, C, D (Experimental): 15 mcg: Sufentanil IV, Sufentanil NanoTab Sublingual, Sufentanil NanoTab Buccal, Sufentanil NanoTab Oral
  Interventions: Drug: Treatment A: Sufentanil IV; Drug: Treatment B: Sufentanil NanoTab Sublingual; Drug: Treatment C: Sufentanil NanoTab Buccal; Drug: Treatment D: Sufentanil NanoTab Oral
- Sequence 2 - Treatment A, B, D, C (Experimental): 15 mcg: IV, Sufentanil NanoTab Sublingual, Sufentanil NanoTab Oral,Sufentanil NanoTab Buccal
  Interventions: Drug: Treatment A: Sufentanil IV; Drug: Treatment B: Sufentanil NanoTab Sublingual; Drug: Treatment C: Sufentanil NanoTab Buccal; Drug: Treatment D: Sufentanil NanoTab Oral
- Sequence 3 - Treatment A, C, B, D (Experimental): 15 mcg: Sufentanil IV, Sufentanil NanoTab Buccal, Sufentanil NanoTab Sublingual, Sufentanil NanoTab Oral
  Interventions: Drug: Treatment A: Sufentanil IV; Drug: Treatment B: Sufentanil NanoTab Sublingual; Drug: Treatment C: Sufentanil NanoTab Buccal; Drug: Treatment D: Sufentanil NanoTab Oral
- Sequence 4 - Treatment A, C, D, B (Experimental): 15 mcg: Sufentanil IV, Sufentanil NanoTab Buccal, Sufentanil NanoTab Oral, Sufentanil NanoTab Sublingual
  Interventions: Drug: Treatment A: Sufentanil IV; Drug: Treatment B: Sufentanil NanoTab Sublingual; Drug: Treatment C: Sufentanil NanoTab Buccal; Drug: Treatment D: Sufentanil NanoTab Oral
- Sequence 5 - Treatment A, D, B, C (Experimental): 15 mcg: Sufentanil IV, Sufentanil NanoTab Oral, Sufentanil NanoTab Sublingual, Sufentanil NanoTab Buccal
  Interventions: Drug: Treatment A: Sufentanil IV; Drug: Treatment B: Sufentanil NanoTab Sublingual; Drug: Treatment C: Sufentanil NanoTab Buccal; Drug: Treatment D: Sufentanil NanoTab Oral
- Sequence 6 - Treatment A, D, C, B (Experimental): 15 mcg: Sufentanil IV, Sufentanil NanoTab Oral, Sufentanil NanoTab Buccal, Sufentanil NanoTab Sublingual
  Interventions: Drug: Treatment A: Sufentanil IV; Drug: Treatment B: Sufentanil NanoTab Sublingual; Drug: Treatment C: Sufentanil NanoTab Buccal; Drug: Treatment D: Sufentanil NanoTab Oral

INTERVENTIONS:
Drug: Treatment A: Sufentanil IV — Sufenta IV (50 mcg/mL) 15 mcg push over 1 minute (IV)
Drug: Treatment B: Sufentanil NanoTab Sublingual — Single Sufentanil NanoTab 15 mcg given sublingually (SL)
Drug: Treatment C: Sufentanil NanoTab Buccal — Treatment C: Single Sufentanil NanoTab 15 mcg given buccally (BU)
Drug: Treatment D: Sufentanil NanoTab Oral — Single Sufentanil NanoTab 15 mcg swallowed (PO)

SUMMARY:
Determine whether the amount of drug absorbed is different if the tablet is placed under the tongue, placed between the cheek and gum, or swallowed.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 18 - 30

Exclusion Criteria:

* pregnant females
* smokers
* pulmonary disease
* sleep apnea

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Palmer, M.D., Study Director — Talphera, Inc
Locations (1):
- PRA, Lenexa, Kansas, United States

REFERENCES:
- [Background] Willsie SK, Evashenk MA, Hamel LG, Hwang SS, Chiang YK, Palmer PP. Pharmacokinetic properties of single- and repeated-dose sufentanil sublingual tablets in healthy volunteers. Clin Ther. 2015 Jan 1;37(1):145-55. doi: 10.1016/j.clinthera.2014.11.001. Epub 2014 Dec 24. PMID 25544247

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Treatment A, B, C, D; Sequence 2: A, B, D, C; Sequence 3: Treatment A, C, B, D; Sequence 4: Treatment A, C, D, B; Sequence Five: Treatments A, D, B, C; Sequence 6: Treatments A, D, C, B: * Treatment A: Sufenta IV (50 mcg/mL) 15 mcg push over 1 minute (IV)
  * Treatment B: Single Sufentanil NanoTab 15 mcg given sublingually (SL)
  * Treatment C: Single Sufentanil NanoTab 15 mcg given buccally (BU)
  * Treatment D: Single Sufentanil NanoTab 15 mcg swallowed (PO)
  A 48-hour washout period will separate each treatment period. The washout begins with the start of dosing.
Period: Overall Study
Arm/Group | Sequence 1: Treatment A, B, C, D | Sequence 2: A, B, D, C | Sequence 3: Treatment A, C, B, D | Sequence 4: Treatment A, C, D, B | Sequence Five: Treatments A, D, B, C | Sequence 6: Treatments A, D, C, B
Started | 4 | 4 | 4 | 5 | 4 | 4
Completed | 3 | 4 | 3 | 4 | 4 | 4
Not Completed | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomly assigned to one of 6 sequences
Groups:
- Treatment A, Followed by Treatment B, C and D in Random Order: Treatment A: Sufenta IV (50 mcg/mL) 15 mcg push over 1 minute (IV) Treatment B: Single Sufentanil NanoTab 15 mcg given sublingually (SL) Treatment C: Single Sufentanil NanoTab 15 mcg given buccally (BU) Treatment D: Single Sufentanil NanoTab 15 mcg swallowed (PO) Sequence 1: A, B, C, D Sequence 2: A, B, D, C Sequence 3: A, C, B, D Sequence 4: A, C, D, B Sequence 5: A, D, B, C Sequence 6: A, D, C, B A 48-hour washout period separated each treatment period. The washout began with the start of dosing.
Arm/Group | Treatment A, Followed by Treatment B, C and D in Random Order
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: AUC (0 - Inf)
Description: total amount of sufentanil absorbed
Time Frame: 24 hours
Population: A The number of subjects (n) in Treatment D was less than the total 22 subjects for the following PK parameters: AUC 0-inf (n=18).
Measure: Mean (Standard Deviation); unit: h.pg/mL
Groups:
- Sufentanil IV: Sufentanil : 15 mcg IV
  PK sampling 0 (predose), 1, 4, 7, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, 720, and 840 minutes and 24 hours after dosing.
- Sufentanil NanoTab Buccal: Sufentanil : 15 mcg buccal
  PK sampling 0 (predose), 10, 20, 30, 40, 50, 60, 70, 80, 90, 120, 180, 240, 360, 480, 600, 720, and 840 minutes and 24 hours after dosing.
- Sufentanil NanoTab Sublingual: Sufentanil : 15 mcg sublingual
  PK sampling 0 (predose), 10, 20, 30, 40, 50, 60, 70, 80, 90, 120, 180, 240, 360, 480, 600, 720, and 840 minutes and 24 hours after dosing.
- Sufentanil NanoTab Oral: Sufentanil : 15 mcg oral
  PK sampling 0 (predose), 10, 20, 30, 40, 50, 60, 70, 80, 90, 120, 180, 240, 360, 480, 600, 720, and 840 minutes and 24 hours after dosing.
Arm/Group | Sufentanil IV | Sufentanil NanoTab Buccal | Sufentanil NanoTab Sublingual | Sufentanil NanoTab Oral
Number analyzed (Participants) | 22 | 22 | 22 | 18
h.pg/mL | 273.8 (61.1) | 212.5 (57.0) | 163.4 (52.5) | 24.9 (14.1)

2. Primary Outcome: Cmax
Description: maximum plasma concentration
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sufentanil IV | Sufentanil NanoTab Buccal | Sufentanil NanoTab Sublingual | Sufentanil NanoTab Oral
Number analyzed (Participants) | 22 | 22 | 22 | 22
pg/mL | 445.1 (312.0) | 58.9 (25.7) | 40.6 (14.8) | 4.3 (3.8)

3. Primary Outcome: Tmax
Description: time to maximum plasma concentration
Time Frame: 24 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Sufentanil IV | Sufentanil NanoTab Buccal | Sufentanil NanoTab Sublingual | Sufentanil NanoTab Oral
Number analyzed (Participants) | 22 | 22 | 22 | 22
hours | 0.07 [0.02 to 0.12] | 0.85 [0.67 to 2.07] | 0.83 [0.33 to 1.50] | 1.11 [0.67 to 3.00]

4. Primary Outcome: CST 1/2
Description: time for maximum plasma concentration to decrease by 50%
Time Frame: 24 hours
Population: The number of subjects (n) in Treatment D was less than the total 22 subjects for the following PK parameters: CST½ (n=16).
Measure: Median (Full Range); unit: hours
Arm/Group | Sufentanil IV | Sufentanil NanoTab Buccal | Sufentanil NanoTab Sublingual | Sufentanil NanoTab Oral
Number analyzed (Participants) | 22 | 22 | 22 | 16
hours | 0.14 [0.05 to 0.68] | 2.28 [0.13 to 4.67] | 2.50 [1.50 to 4.83] | 2.00 [0.83 to 4.67]

ADVERSE EVENTS:
Groups:
- Sufentanil IV: Sufentanil : 15 mcg IV
- Sufentanil NanoTab Buccal: Sufentanil : 15 mcg buccal
- Sufentanil NanoTab Sublingual: Sufentanil : 15 mcg sublingaul
- Sufentanil NanoTab Oral: Sufentanil : 15 mcg oral
Arm/Group | Sufentanil IV | Sufentanil NanoTab Buccal | Sufentanil NanoTab Sublingual | Sufentanil NanoTab Oral
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 8/25 | 4/24 | 5/24 | 3/23
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil IV (N=25) | Sufentanil NanoTab Buccal (N=24) | Sufentanil NanoTab Sublingual (N=24) | Sufentanil NanoTab Oral (N=23)
nausea (Gastrointestinal disorders) | 4 | 1 | 0 | 2
headache (Nervous system disorders) | 2 | 2 | 1 | 0
photophobia (Eye disorders) | 1 | 0 | 0 | 0 — all subjects received naltrexone 50 mg BID
abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
fatigue (General disorders) | 0 | 0 | 1 | 0
decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
flat effect (Psychiatric disorders) | 1 | 1 | 1 | 0
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
infusion site pain (General disorders) | 1 | 0 | 0 | 0
dizziness (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
requires prior approval